CLINICAL TRIAL: NCT02157662
Title: Coronary Atherosclerosis in Outlier Subjects: Protective and Individual Risk Factor Evaluation
Brief Title: GISSI Outliers CAPIRE
Acronym: CAPIRE
Status: Completed | Type: Observational
Sponsor: Gruppo di Ricerca GISSI (Other)
Responsible Party: Sponsor
Other Study IDs: K10
Record Dates: First submitted 2014-05-27; First posted 2014-06-06 (Estimated); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood and serum. Lipid profile Metabolic profile (HbA1c, HOMA index) inflammatory profile (CRP, LP-PLA, pentraxine 3, MCP-1, IL-8, IL-10, IL-5, P-selectin, ICAM, VCAM-1, CD40L, TIMP-1, MMP Genetic profile: chromosome polymorphism 9 (9p21)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- No coronary disease and risk factors >=3
- Coronary disease and risk factors 0-1: Diffuse coronary atherosclerosis extended to more than 5 of the 16 segments according to the American Heart Association classification38 and 0-1 risk factor (reported by the subject or documented at the MDCT) with the exclusion of patients with type 1 or type 2 diabetes mellitus as single risk factor.
- No coronary disease and risk factors 0-1
- Coronary disease and risk factors >=3: Subjects with diffuse coronary atherosclerosis extended to more than 5 of the 16 segments according to the American Heart Association classification38 and 3 or more risk factors (reported by the subject or documented at the MDCT) with the exclusion of patients with type 1 or type 2 diabetes mellitus as single risk factor

SUMMARY:
The risk of developing clinical manifestations of ischemic heart disease is currently assessed by using integrated multifactorial prediction models based on the presence of non-modifiable risk factors, such as age, gender and a family history of early ischemic heart disease along with risk factors which are defined as conventional, such as arterial hypertension, hypercholesterolemia, cigarette smoking and diabetes mellitus.

However, if the relationship between risk factors and ischemic heart disease clinical manifestations shows some limitations, the relation between risk factors and the coronary atherosclerosis process underlying most ischemic syndromes seems to be even weaker.

In fact there is significant individual variability and the limits of such relationship are demonstrated by a non negligible number of subjects at the outliers of mean behaviour of the prediction model. At one outlier, in the presence of multiple risk factors, these subjects do not develop neither coronary events nor coronary atherosclerosis whereas, at the other, coronary events and disease occur in the absence of risk factors.This study aims at detecting new protection and susceptibility factors, thus enabling to formulate new etiopathogenetic hypotheses concerning coronary atherosclerosis and to identify new therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Group A: subjects with total absence of coronary atherosclerosis and 3 or more risk factors (reported by the subject or documented at the MDCT)
* Group B: subjects with diffuse coronary atherosclerosis extended to more than 5 of the 16 segments according to the American Heart Association classification and 0-1 risk factor (reported by the subject or documented at the MDCT) with the exclusion of patients with type 1 or type 2 diabetes mellitus as single risk factor.

Using the same criteria, two control populations will be selected, with a case:control 1:1 ratio, consisting in:

* Group C: subjects with total absence of coronary atherosclerosis and 0-1 risk factor (reported by the subject or documented at the MDCT)
* Group D: subjects with diffuse coronary atherosclerosis extended to more than 5 of the 16 segments according to the American Heart Association classification and 3 or more risk factors (reported by the subject or documented at the MDCT) with the exclusion of patients with type 1 or type 2 diabetes mellitus as single risk factor.

Exclusion Criteria:

* common contraindications to MDCT (chronic renal failure with serum creatinine > 2.0 mg/dl, suspected pregnancy, arrhythmias, body mass index > 40, allergy to iodized contrast agent).
* previous cardiovascular events (heart failure, acute myocardial infarction, unstable angina, chronic stable angina, previous percutaneous or surgery coronary revascularization) both clinically evident and found by conventional diagnostic methods previous performed.
* subjects which MDCT does not meet the quality control criteria defined below in the protocol.
* patients with previous documented or identified at the moment of MDCT such as dilated cardiomyopathy regardless of etiology, obstructive hypertrophic cardiomyopathy, atrial fibrillation, myocarditis and inflammatory vascular disease.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female subjects between 45 and 75 years old who, in the absence of any previous clinical manifestations of ischemic heart disease, will undergo coronary arteries study.
Sampling Method: Probability Sample
Enrollment: 544 (Actual)
Dates: Start 2011-01; Primary Completion 2013-07 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Number of patients in each Group with a cardiovascular Event | 5 years

SECONDARY OUTCOMES:
Polymorphisms associated with chromosome 9 in each patient | At enrollment visit

CONTACTS AND LOCATIONS:
Locations (10):
- Italy (9):
  - Nuovo Ospedale Versilia - SC Cardiologia, Lido di Camaiore, Lucca
  - Ospedale Santa Croce - U.O.C. Cardiologia, Fano, PU
  - Ospedale Civile Augusto Murri - U.O. Cardiologia, Fermo
  - IFC CNR - Ospedale Pasquinucci - U.O. Cardiologia Adulti, Massa
  - Ospedale Policlinico - Divisione di Cardiologia, Modena
  - Az. Ospedaliera Universitaria di Parma - U.O. Cardiologia, Parma
  - Azienda Ospedaliero Universitaria Pisana - U.O. Radiodiagnostica I, Pisa
  - IFC CNR Fondazione Toscana G. Monasterio - S.A. Emodinamica, Pisa
  - AOU Santa Maria della Misericordia - Angiografia e Radiologia Interventistica, Udine
- Cardiocentro Ticino - SRC, Lugano, Switzerland

REFERENCES:
- [Background] Magnoni M, Andreini D, Gorini M, Moccetti T, Modena MG, Canestrari M, Berti S, Casolo G, Gabrielli D, Marraccini P, Pontone G, Masson S, Latini R, Maggioni AP, Maseri A; CAPIRE Study Group. Coronary atherosclerosis in outlier subjects at the opposite extremes of traditional risk factors: Rationale and preliminary results of the Coronary Atherosclerosis in outlier subjects: Protective and novel Individual Risk factors Evaluation (CAPIRE) study. Am Heart J. 2016 Mar;173:18-26. doi: 10.1016/j.ahj.2015.11.017. Epub 2015 Dec 17. PMID 26920592
- [Background] Magnoni M, Masson S, Andreini D, Moccetti T, Modena MG, Canestrari M, Berti S, Casolo G, Gabrielli D, Marraccini P, Pontone G, Latini R, Maggioni AP, Maseri A; CAPIRE Study Group. Usefulness of High-Sensitivity Cardiac Troponin T for the Identification of Outlier Patients With Diffuse Coronary Atherosclerosis and Low-Risk Factors. Am J Cardiol. 2016 May 1;117(9):1397-404. doi: 10.1016/j.amjcard.2016.02.002. Epub 2016 Feb 17. PMID 26976791
- [Background] Andreini D, Magnoni M, Conte E, Masson S, Mushtaq S, Berti S, Canestrari M, Casolo G, Gabrielli D, Latini R, Marraccini P, Moccetti T, Modena MG, Pontone G, Gorini M, Maggioni AP, Maseri A; CAPIRE Investigators. Coronary Plaque Features on CTA Can Identify Patients at Increased Risk of Cardiovascular Events. JACC Cardiovasc Imaging. 2020 Aug;13(8):1704-1717. doi: 10.1016/j.jcmg.2019.06.019. Epub 2019 Aug 14. PMID 31422137
- [Background] Ferrannini G, Manca ML, Magnoni M, Andreotti F, Andreini D, Latini R, Maseri A, Maggioni AP, Ostroff RM, Williams SA, Ferrannini E. Coronary Artery Disease and Type 2 Diabetes: A Proteomic Study. Diabetes Care. 2020 Apr;43(4):843-851. doi: 10.2337/dc19-1902. Epub 2020 Jan 27. PMID 31988066
- [Background] Conte E, Andreini D, Magnoni M, Masson S, Mushtaq S, Berti S, Canestrari M, Casolo G, Gabrielli D, Latini R, Marraccini P, Moccetti T, Modena MG, Pontone G, Gorini M, Maggioni AP, Maseri A; CAPIRE Investigators, Steering Committee; Imaging Core Laboratory; Centralized biobank and biomarker core laboratory; Central ECG Reading; Psychologists CRF Group; Participating Centers and Investigators. Association of high-risk coronary atherosclerosis at CCTA with clinical and circulating biomarkers: Insight from CAPIRE study. J Cardiovasc Comput Tomogr. 2021 Jan-Feb;15(1):73-80. doi: 10.1016/j.jcct.2020.03.005. Epub 2020 Jun 11. PMID 32563713
- [Derived] Magnoni M, Andreini D, Andreotti F, Latini R, Maseri A, Nicoletti A, Maggioni AP, Caligiuri G. Leukocyte-shed soluble CD31 unmasks coronary disease in low-risk outliers and provides source-specific inflammatory signatures of vulnerable plaques. Atherosclerosis. 2025 Aug;407:120410. doi: 10.1016/j.atherosclerosis.2025.120410. Epub 2025 Jun 13. PMID 40543300
- [Derived] Ferrannini E, Manca ML, Ferrannini G, Andreotti F, Andreini D, Latini R, Magnoni M, Williams SA, Maseri A, Maggioni AP. Differential Proteomics of Cardiovascular Risk and Coronary Artery Disease in Humans. Front Cardiovasc Med. 2022 Feb 4;8:790289. doi: 10.3389/fcvm.2021.790289. eCollection 2021. PMID 35187107